CLINICAL TRIAL: NCT03667456
Title: Evaluation of the Uses of a Digital-assisted Self-rehabilitation Device Coupled With a Tele-reeducative Follow-up in Patients With Parkinson's Disease on a Defined Health Area (TELE-PARK)
Brief Title: Evaluation of the Uses of a Digital-assisted Self-rehabilitation Device (TELE-PARK)
Acronym: TELE-PARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Collaborators: Réseau Parkinson Bretagne (Unknown); Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A02379-44
Record Dates: First submitted 2018-08-17; First posted 2018-09-12 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2019-11

CONDITIONS: Parkinson Disease; Parkinson's Syndrome
Keywords: Parkinson; Serious Game; Self management; Rehabilitation; Telemedicine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-rehabilitation by digital support (Experimental): Provision to patients selected by doctors or physiotherapists of an interactive digital tool (tablet + inertial sensor) to support self-rehabilitation home Parkinson's patients.
  Monitoring and regulation of remote self-reeducation by tele-reeducation. Evaluation of the acceptance of the tool and the quality of life of the patients by questionnaire at day 0, and two and twelve months after.
  Interventions: Procedure: Self-rehabilitation by digital support

INTERVENTIONS:
Procedure: Self-rehabilitation by digital support — Provision to patients selected by doctors or physiotherapists of an interactive digital tool (tablet + inertial sensor) to support self-rehabilitation home Parkinson's patients.

SUMMARY:
Evaluate the use by the patient and his family and professional environment of a self-rehabilitation device with follow-up in tele-rehabilitation in people with Parkinson's disease taking into account the different actors within a health area (health professionals and paramedics in structure and in liberal).

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Men and women over the age of 18
* With Parkinson's syndrome due to idiopathic Parkinson's disease or related syndromes
* Presenting a complaint about balance and/or walking
* With possible walking over a perimeter of at least 100 meters with or without technical aid
* Hoehn and Yahr scale < or = to 4
* Formulating their free and informed consent in writing.

Health professionals:

- physiotherapists and physiatrists hospital or voluntary volunteers practicing in the territory of health 5 in Brittany agreeing to participate in the study

Exclusion Criteria:

* Orthopedic and rheumatologic pathologies that may prevent the achievement of measures
* Comprehension disorders preventing the implementation of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
UTAUT Questionnaire | 12 months
  Questionnaire of acceptability / acceptance of the tool and its use by professionals based on the Unified Theory of Acceptance and Use Technology (UTAUT).

SECONDARY OUTCOMES:
UTAUT Questionnaire | 12 months
  Questionnaires for integrating the tool and its use at 12 months for professionals and patients / entourage
Observance | 12 months
  Observance of self-rehabilitation using tablet data at 2 months and 12 months: the tablet records the number of sessions performed, their duration, the number and type of exercises performed
SF36 | 12 months
  The 36-Item Short Form Health Survey is assessing the subjective quality of life of patients summarized in two component summary scores, the Physical Component Summary (PCS) and the Mental Component Summary (MCS) scores. The SF-36 includes one multi-item scale that assesses eight health concepts. All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible. Aggregate scores are compiled as a percentage of the total points possible, using the RAND scoring table. The scores from those questions that address each specific area of functional health status are then averaged together, for a final score within each of the 8 dimensions measured. Reliability is measured by Cronbach's alpha coefficient. Its value is less than or equal to 1. It is considered "acceptable" from 0.7.
Rosenberg SES | 12 months
  Rosenberg's self-esteem scale (SES) assesses self-esteem. The questionnaire consists of 10 items of which 5 evaluate positive self-esteem and 5 negative self-esteem. The answer varies according to a four-point Likert-type scale from "Strongly disagree" (1) to "Totally agree" (4). A score between 10 and 40 is obtained. A score below 25 means very low self-esteem; a score between 25 and 31 means low self-esteem; a score between 31 and 34 means an average self-esteem; a score between 34 and 39 means a strong self-esteem; a score above 39 means a very strong self-esteem.
Zarit's Score | 12 months
  The Zarit scale assesses the emotional, physical and financial burden for caregivers of caring for someone with a loss of autonomy. The 22-item grid allows an assessment of this burden, ranging from mild to moderate to severe. The total score (sum of the 22-item scores) ranges from 0 to 88.
  A score less than or equal to 20 indicates a low or no burden; a score between 21 and 40 indicates a light burden; a score between 41 and 60 indicates a moderate burden; a score above 60 indicates a severe burden
Performance indicators | 12 months
  Alternatives that would have been implemented to meet the difficulties of the liberal therapist with his patient, number of kilometers saved by telereducation
VAS Satisfaction | 12 months
  The Visual Analogue Scale (VAS) allows a quick estimate of the level of satisfaction of patients by positioning themselves on a line whose extremities indicate the lowest level on the left (0) and the strongest on the right (10)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gallien, Doctor, Study Director — Pole Saint Hélier
Locations (1):
- Pôle Saint Hélier, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No